CLINICAL TRIAL: NCT03863782
Title: Lyon Sarcoid Uveitis Cohort
Acronym: LUCS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2018_001
Record Dates: First submitted 2018-05-17; First posted 2019-03-05 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Sarcoid Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoid uveitis: The cohort is composed by patients diagnosed or treated for sarcoid uveitis in the departement for Internal Medicine, Croix Rousse Hospital, Lyon, France.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No specific intervention. Collection of clinical data

SUMMARY:
Sarcoidosis is a systemic disease with unknown etiology. Chronicity of the disease is observed in 1/3 of cases. Five percent of the affected patients are expected to die due to pulmonary worsening. After pulmonary complications, ocular complications are one of the most frequent complications. In hospital setting 2 to 15% of patients who come for initial uveitis diagnosis are after examination due to Sarcoidosis. Sarcoidosis diagnosis is based on paraclinical exams (biological, radiography) and histological confirmation. Corticotherapy (local or general) is usually used to cure sarcoid uveitis. In case of failure immunosuppressor or anti-tumor necrosis factor (TNF) can be used. In 10% of cases ocular symptoms including blindness are observed. Only treatment administrated quickly after diagnosis of sarcoid uveitis can prevent from ophthalmologic complications.

The main objective of the Lyon Sarcoid Uveitis Cohort study is to analyze the relevance of the paraclinical exam for sarcoid uveitis diagnosis, and to define a better visual and extra-ophthalmologic prognosis and describe the therapeutic practice in our Department.

This study is proposed to all patients diagnosed with Sarcoid uveitis with a histological confirmation and referred to the internal medicine department of the Croix-Rousse hospital, Lyon, France, for etiologic diagnosis or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoid uveitis
* First consultation in the department of Internal Medicine at the Croix-Rousse hospital, Lyon, France

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is proposed to all patients with a diagnosis of sarcoid uveitis and referred to the Internal Medicine department of the Croix-Rousse hospital
  .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution (persistence or resolution) evaluated by gradation of SEN | At one year after diagnosis
  Persistence of disease is characterized by persistence of intraocular inflammation evaluated by gradation of SEN. (reference: A Standardization Grading System for Scleritis . Ophthalmology 2011 Apr;118(4):768-71). SEN score ranges from 0 to 5 (resolution = score 0 and persistence = score >0)

SECONDARY OUTCOMES:
Anatomic characteristic of sarcoid uveitis | At inclusion visit
  The anatomic characteristics of sarcoid uveitis will be described: anterior or posterior inflammation of greater rings of iris, ciliary margin of iris
Corticoid treatment duration | At one year after diagnosis
  Treatment used to cure uveitis: duration of corticotherapy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danjou W, Pradat P, Jamilloux Y, Gerfaud-Valentin M, Kodjikian L, Trad S, Seve P. Usefulness of the QuantiFERON test for the diagnosis of tubercular uveitis and the predictions of response to antituberculosis treatment. Br J Ophthalmol. 2023 Apr;107(4):500-504. doi: 10.1136/bjophthalmol-2021-318868. Epub 2021 Oct 28. PMID 34711577
- [Derived] Cotte P, Pradat P, Kodjikian L, Jamilloux Y, Seve P. Diagnostic value of lymphopaenia and elevated serum ACE in patients with uveitis. Br J Ophthalmol. 2021 Oct;105(10):1399-1404. doi: 10.1136/bjophthalmol-2020-316563. Epub 2020 Sep 11. PMID 32917626